CLINICAL TRIAL: NCT06822205
Title: Identification and Treatment of Renal Stenosis in Transplanted Kidneys
Acronym: TRAS
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: TRAS
Record Dates: First submitted 2024-11-28; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-11

CONDITIONS: Renal Artery Stenosis
MeSH Terms: conditions — Renal Artery Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Renal artery stenosis is a complication that may follow kidney transplantation1-5. Renal artery stenosis greater than 50% of the lumen of the artery, associated with clinical symptoms or laboratory worsening of renal function, may lead to transplant failure, however, the indications for treatment and the modalities of treatment remain, to date, a debated topic in the literature. The guidelines of the European Society of Urology recommend endovascular treatment as the first-line treatment by means of angioplasty and/or stent placement6. A recent review of the literature7 examined the results of 56 studies: the results fully support endovascular treatment of the disease which appears to be effective and with a low rate of complications.

DETAILED DESCRIPTION:
The primary objectives of the study are to evaluate the efficacy (in terms of technical success and graft salvage) and safety (in terms of complications) of endovascular treatment using stenting in patients with renal artery stenosis following kidney transplantation.

Patients undergoing endovascular treatment of renal stenosis following kidney transplantation at the Vascular Surgery Unit from January 2020 to April 2023 (retrospective phase) and from May 2023 up to 2 years from the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Indication of renal transplant and diagnosis of renal artery stenosis of the transplant
* Obtaining informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing endovascular treatment of renal stenosis following kidney transplantation at the Vascular Surgery Unit from January 2020 to April 2023 (retrospective phase) and from May 2023 up to 2 years from the start of the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of stenosis | From the first patient enrolled up to the 30th patient, an average of 3 years
  Efficacy is assessed by a reduction in stenosis of at least 50% based on the TC image
Renal function improvement | From the first patient enrolled, up to the 30th patient. An average of 3 years
  It is assessed through the improvement in eGFR and Creatinine values, compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Gargiulo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS AOU di Bologna Policlinico di Sant'Orsola, Bologna, Italy